CLINICAL TRIAL: NCT05561270
Title: Investigation of Light Exposure on Pain Severity and Quality of Life in Individuals With Hypermobile Ehlers-Danlos Syndrome: A Pilot Study
Brief Title: Light Exposure on Pain in Hypermobile Ehlers-Danlos Syndrome
Acronym: LEEDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BHS-1755
Record Dates: First submitted 2022-09-20; First posted 2022-09-30 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Ehlers-Danlos Syndrome; Pain, Chronic
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Single-center, randomized clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- White LED light (Sham Comparator): Exposure to white LED light for 1-2 hours/day x 10 weeks
  Interventions: Device: White LED light
- Green LED light (Experimental): Exposure to green LED light for 1-2 hours/day x 10 weeks
  Interventions: Device: Green LED light

INTERVENTIONS:
Device: White LED light — Exposure to white LED light for 1-2 hours/day x 10 weeks
  Arms: White LED light
Device: Green LED light — Exposure to green LED light for 1-2 hours/day x 10 weeks
  Arms: Green LED light

SUMMARY:
Chronic pain is a major complaint among many individuals living with hypermobile Ehlers Danlos Syndrome (hEDS) and may have a severe impact on quality of life and activities of daily living. Given the complexity of the disease's pathophysiology, effective treatments are limited. This investigation will examine the impacts of green light exposure on subject-reported pain severity and symptoms. Knowing whether this intervention can improve pain and quality of life in this population may offer valuable guidance to clinicians who treat hEDS patients and to hEDS patients themselves.

DETAILED DESCRIPTION:
Chronic pain is a major complaint among many individuals living with hEDS and may have a severe impact on quality of life and activities of daily living. Given the complexity of the disease's pathophysiology, effective treatments are limited. A multidisciplinary approach, including pharmacologic and nonpharmacologic pain management, physical therapy, occupational therapy, and psychological treatment alongside prophylactic care and interventions has been recommended for these patients. The application of light for pain and injury has been studied for some time. More recently, specific colored light has shown promise in treating chronic pain. Green light emitting diodes significantly reduced the number of headache days in people with episodic migraine or chronic migraine. Additionally, green light emitting diodes significantly improved multiple secondary outcome measures including quality of life and intensity and duration of the headache attacks. As no adverse events were reported, green light emitting diodes may provide a treatment option for those patients who prefer non-pharmacological therapies or may be considered in complementing other treatment strategies. This investigation will examine the impacts of green light exposure on subject-reported pain severity and symptoms. Knowing whether this intervention can improve pain and quality of life in this population may offer valuable guidance to clinicians who treat hEDS patients and to hEDS patients themselves.

Subjects will be enrolled for a total of 10 weeks, inclusive of either a 10-week control white light exposure period or a 10-week experimental green light exposure period. Central sensitization inventory will be used to determine the degree of central sensitization contributing to pain for each subject at baseline.

All subjects will be provided with a light source that will achieve light intensity of 4 and 100 lux measured at approximately 1 and 2 meters from point of exposure from a lux meter to determine the illuminance and luminous emittance of the LED strips. Subjects will be free to change the distance of the light source between 1 and 2 meters from their eyes to find the intensity that best suited them. The equipment will be provided during the initial clinic visit or mailed to the patients' homes and they will be instructed to use it in a dark room with no other source of light, except provided source, for a minimum of 1 hour every day, with the option to increase the exposure time to 2 hours daily for 10 weeks. The subjects will be asked to eliminate other sources of extraneous light (no use of televisions, computers, or smartphones; curtains drawn and existing room lights turned off) and will be encouraged to keep their eyes open, to blink at a normal rate, and not to stare directly at the light source. Subjects will be encouraged to engage in any activity while undergoing light exposure, such as reading or listening to music, and avoid falling asleep. Subjects will have the option to receive a daily text message/email reminder about light exposure and questionnaire completion. They will be provided with questionnaires to document the primary and secondary outcomes. Subjects will be allowed to continue their current medical therapy as recommended by their treating physicians. They will also be allowed to start any new medications as recommended by their treating physicians and instructed to document all medications used for their pain. Subjects will self-report the light exposure log, pain medication log, and pain severity data daily to minimize the chances of recall bias. Short-Form McGill Pain Questionnaire (SFMPQ) will be self-reported by subjects every 2 weeks. Short-Form 36 Health Survey (SF-36) data will be self-reported by subjects at their initial visit, 5-week visit, and 10-week visit. Athens Insomnia Scale (AIS) and Test My Brain (TMB) cognitive performance measures will be completed at baseline and week 10. The daily log and McGill Short-Form will be completed on paper. Other measures will be set up electronically for ease of patient completion and submission, but paper evaluations will be available as a back-up if there are technological difficulties. The TMB cognitive performance tests are performed on a computerized interactive interface and patients will be given access to the activities.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older and able to speak, read, and understand English
2. Diagnosed with hEDS
3. Average numeric pain score of 5 out of 10 or greater over the 10 weeks prior to enrolling in the study and failure of medical therapy to control the pain

Exclusion Criteria:

1. Initiation of any new analgesic therapy within 30 days of enrollment (note: chronic therapy with a stable regimen maintained for at least 30 days prior to enrollment is permitted)
2. Serious mental illness, defined as distortions of perception, delusions, hallucinations, and unusual behaviors resulting in loss of contact with reality or Major Depression Disorder
3. History of color blindness or uncorrected cataracts
4. Receiving remuneration, or litigation pending, for their medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Changes in pain intensity as measured by subject-reported numeric pain severity (NPS) rating | 10 weeks
  Subjects will report pain intensity daily as a numeric pain severity (NPS) rating, a subjective pain scale ranging from 0 (no pain) to 10 (most severe pain)

SECONDARY OUTCOMES:
Qualitative changes in pain as measured by Short-Form McGill Pain Questionnaire (SFMPQ) | 10 weeks
  Subjects will describe pain per Short-Form McGill Pain Questionnaire (SFMPQ) every 2 weeks through the duration of their participation. In this questionnaire, subjects will rate their pain on scales from 0 (no pain) to 3 (severe pain). Higher scores indicate worse outcomes.
Changes in frequency of pain medication usage | 10 weeks
  Subjects will report frequency of any pain medications used through the duration of their participation
Changes in dosage of pain medication used | 10 weeks
  Subjects will report dosages of any pain medications used through the duration of their participation
Health-related quality of life as measured by subject-reported Short-Form 36 Health Survey (SF-36) | 10 weeks
  Subjects will complete Short-Form 36 Health Survey (SF-36) at baseline, week 5, and week 10. This survey asks subjects to qualitatively rate their health-related limitations of activities of daily living on Likert scales (e.g. ranging from "no limitation" to "severe limitation").
Insomnia as measured by subject-reported Athens Insomnia Scale | 10 weeks
  Subjects will complete Athens Insomnia Scale at baseline and week 10. Subjects will rate aspects of their sleep quality on this scale from 0 (no problem) to 3 (severe problem).
Verbal memory as measured by "Test My Brain" (TMB) digital neuropsychiatry cognitive performance test | 10 weeks
  Subjects will complete "Test My Brain" (TMB) digital neuropsychiatry cognitive performance test assessing verbal memory at baseline and week 10. This computerized test calculates the subject's performance in learning and recognizing sets of word pairs. Performance is digitally analyzed, quantified and compared against normative data by age, gender and education level. Higher scores are associated with improved outcomes.
Sustained attention as measured by "Test My Brain" (TMB) digital neuropsychiatry cognitive performance test | 10 weeks
  Subjects will complete "Test My Brain" (TMB) digital neuropsychiatry cognitive performance test assessing sustained attention at baseline and week 10. This computerized test calculates the subject's performance in recognizing and responding to sets of rapidly transitioning images. Performance is digitally analyzed, quantified and compared against normative data by age, gender and education level. Higher scores are associated with improved outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Noto, DO, Principal Investigator — NYITCOM
Locations (1):
- New York Institute of Technology College of Osteopathic Medicine, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Syx D, De Wandele I, Rombaut L, Malfait F. Hypermobility, the Ehlers-Danlos syndromes and chronic pain. Clin Exp Rheumatol. 2017 Sep-Oct;35 Suppl 107(5):116-122. Epub 2017 Sep 28. PMID 28967365
- [Background] Hakimi A, Bergoin C, Mucci P. What are the most important symptoms to assess in hypermobile Ehlers-Danlos syndrome? A questionnaire study based on the Delphi technique. Disabil Rehabil. 2022 Dec;44(26):8325-8331. doi: 10.1080/09638288.2021.2012839. Epub 2021 Dec 18. PMID 34927503
- [Background] Cheng K, Martin LF, Slepian MJ, Patwardhan AM, Ibrahim MM. Mechanisms and Pathways of Pain Photobiomodulation: A Narrative Review. J Pain. 2021 Jul;22(7):763-777. doi: 10.1016/j.jpain.2021.02.005. Epub 2021 Feb 23. PMID 33636371
- [Background] Martin LF, Patwardhan AM, Jain SV, Salloum MM, Freeman J, Khanna R, Gannala P, Goel V, Jones-MacFarland FN, Killgore WD, Porreca F, Ibrahim MM. Evaluation of green light exposure on headache frequency and quality of life in migraine patients: A preliminary one-way cross-over clinical trial. Cephalalgia. 2021 Feb;41(2):135-147. doi: 10.1177/0333102420956711. Epub 2020 Sep 9. PMID 32903062
- [Background] Martin L, Porreca F, Mata EI, Salloum M, Goel V, Gunnala P, Killgore WDS, Jain S, Jones-MacFarland FN, Khanna R, Patwardhan A, Ibrahim MM. Green Light Exposure Improves Pain and Quality of Life in Fibromyalgia Patients: A Preliminary One-Way Crossover Clinical Trial. Pain Med. 2021 Feb 4;22(1):118-130. doi: 10.1093/pm/pnaa329. PMID 33155057